CLINICAL TRIAL: NCT01742611
Title: ASP1585 Phase 3 Long-term Study in Chronic Kidney Disease Patients With Hyperphosphatemia Not on Dialysis
Brief Title: Long-term Study in Chronic Kidney Disease Patients With Hyperphosphatemia Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1585-CL-0102
Record Dates: First submitted 2012-12-04; First posted 2012-12-05 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Kidney Disease; Renal Insufficiency; Hyperphosphatemia
Keywords: CKD; Not on dialysis; ASP1585; Bixalomer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Hyperphosphatemia | interventions — bixalomer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP1585 group (Experimental)
  Interventions: Drug: ASP1585

INTERVENTIONS:
Drug: ASP1585 — oral
  Other Names: LY101; AMG223; bixalomer

SUMMARY:
This is a multi-center, open-labeled, non-comparative study to examine the safety and efficacy of ASP1585 for long-term dosing in chronic kidney disease patients with hyperphosphatemia not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed study 1585-CL-0101 or new patients who meet following criteria
* Chronic kidney disease patients (eGFR < 60 mL/min/1.73 m2)
* Serum phosphorus measurement ≧4.6 mg/dl, <9.0 mg/dl
* Written informed consent

Exclusion Criteria:

* Patients with gastrointestinal surgery or enterectomy
* Patients with severe cardiac diseases
* Patients with severe constipation or diarrhea
* Patients with a history or complication of malignant tumors
* Patients with uncontrolled hypertension
* Patients treated with parathyroid intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time-course changes in serum phosphorus levels | During 48 week treatment

SECONDARY OUTCOMES:
Achievement rate of the target range of serum phosphorus level | During 48 week treatment
Time to achieve the target range of serum phosphorus level | During 48 week treatment
Time-course changes in serum calcium levels | During 48 week treatment
Time-course changes in serum intact PTH (parathyroid hormone) levels | During 48 week treatment
Safety assessed by the incidence of adverse events, vital signs, labo-tests and 12-lead ECGs | During 48 week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu